CLINICAL TRIAL: NCT07094204
Title: A Phase 1 Study of ASP5834 in Participants With Locally Advanced (Unresectable) or Metastatic Solid Tumor Malignancies With KRAS Mutations or KRAS Amplifications
Brief Title: A Study to Find a Suitable Dose of ASP5834 in Adults With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5834-CL-1001; 2025-522082-29-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor; Non-Small-Cell Lung Cancer; Pancreatic Ductal Adenocarcinoma; Colorectal Cancer
Keywords: Solid Tumor; Cancer; Malignancy; Metastasis; Pharmacokinetics; ASP5834; KRAS G12V; KRAS G12D; KRAS G12C; KRAS G12R; KRAS G12A; KRAS G13D; CRC; NSCLC; PDAC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ASP5834 Dose Escalation (Experimental): Participants will receive sequential doses levels of ASP5834 intravenously following 1 of 2 dose regimens.
  Interventions: Drug: ASP5834
- ASP5834 Dose Expansion (Tumor/ Mutation Specific) (Experimental): Participants with select tumor types will receive 1 of 2 dose regimens of ASP5834 with dose level(s) selected from dose escalation.
  Interventions: Drug: ASP5834
- ASP5834 Dose Expansion (Dose-ranging) (Experimental): Participants will receive dose level(s) and regimen of ASP5834 based on emerging data from Dose Escalation alone or Dose Escalation and Dose Expansion cohorts.
  Interventions: Drug: ASP5834
- ASP5834 combination therapy Dose Escalation (Experimental): Participants will receive sequential doses levels of ASP5834 intravenously following 1 of 2 dose regimens based on emerging data. Panitumumab will be administered every 2 weeks.
  Interventions: Drug: ASP5834; Drug: panitumumab
- ASP5834 monotherapy therapy Dose Expansion (Experimental): Participants will receive 1 of 2 dose regimens of ASP5834.
  Interventions: Drug: ASP5834
- ASP5834 combination therapy Dose Expansion (Experimental): Participants will receive ASP5834 and panitumumab with dose level(s) and regimen selected from dose escalation (Combination Therapy). Panitumumab will be administered every 2 weeks.
  Interventions: Drug: ASP5834; Drug: panitumumab

INTERVENTIONS:
Drug: ASP5834 — Intravenous infusion
Drug: panitumumab — Intravenous infusion
  Arms: ASP5834 combination therapy Dose Escalation; ASP5834 combination therapy Dose Expansion

SUMMARY:
Genes contain genetic code which tell the body which proteins to make. Many types of cancer are caused by changes, or mutations, in a gene called KRAS. Researchers are looking for ways to stop the actions of abnormal proteins made from the mutated KRAS gene.

ASP5834 is being studied in people with solid tumors who have certain KRAS gene mutations. Some people with solid tumors of the colon or rectum (colorectal cancer), will be given ASP5834 with panitumumab. Panitumumab is a treatment for colorectal cancer. In this study, the researchers will learn how ASP5834 is processed by and acts upon the body. This information will help find a suitable dose of ASP5834 and check for any potential medical problems from the treatment.

The main aims of this study are to check the safety of ASP5834 given by itself or given with panitumumab, and how well it is tolerated; and to find a suitable dose of ASP5834 given by itself or given with panitumumab.

People in this study will be adults with locally advanced, unresectable, or metastatic solid tumors with certain KRAS gene mutations. Locally advanced means the cancer has spread to nearby tissue. Unresectable means the cancer cannot be removed by surgery. Metastatic means the cancer has spread to other parts of the body. The key reasons people cannot take part are if they have specific uncontrollable cancers such as symptomatic or untreated cancers in nervous system, or have a specific heart condition, or infections.

In this study, ASP5834 is being given to humans for the first time. This is an open-label study. This means that people in this study and clinic staff will know that they will receive ASP5834 by itself or ASP5834 with panitumumab.

This study will be in 2 parts:

Part 1 is called Dose Escalation. Different small groups of people will receive lower to higher doses of either: ASP5834 by itself or ASP5834 with panitumumab. Only people who have colorectal cancer will receive ASP5834 with panitumumab. People with any type of solid tumor will receive ASP5834 by itself. For each dose, all medical problems will be recorded. A medical expert panel will check the results and decide if the next group can receive a higher dose of ASP5834. The panel will do this until the planned maximum number of people are treated or until suitable doses have been selected for Part 2.

Part 2 is called Dose Expansion. Other different small groups of people will receive ASP5834 or ASP5834 with panitumumab. They will receive the most suitable doses worked out from Part 1.

In both parts of the study, the study treatments ASP5834 and panitumumab will be given through a vein. This is called an infusion. Each study treatment cycle is either 21 days or 28 days long. People will continue study treatment until: they have medical problems from the study treatment they can't tolerate; their cancer gets worse; they start other cancer treatment; or they ask to stop study treatment.

People will visit the clinic on certain days during their study treatment, with extra visits during the first 2 cycles of study treatment. The study doctors will check for any medical problems from ASP5834. Also, people in the study will have a health check. On some visits they will also have scans to check for any changes in their cancer. Tumor samples will be taken at certain visits during study treatment with the option of a tumor sample being taken if people's cancer gets worse or the cancer comes back.

People will visit the clinic shortly after stopping treatment for a health check. After this, people will have health checks every couple of months to check the condition of their cancer. The number of visits and checks done will depend on the health of each person and whether they completed their study treatment or not. It is expected that people will be in this study for about 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically confirmed locally advanced (unresectable) or metastatic solid tumor malignancy with a documented Kirsten rat sarcoma viral oncogene homolog (KRAS) G12V, G12D, G12C, G12R, G12A or G13D mutation or KRAS amplification (copy number >/= 4) determined by local testing.

  * For a participant with a documented KRAS amplification, only those with no other co-occurring KRAS mutation or those with a co-occurring KRAS G12V, G12D, G12C, G12R, G12A or G13D mutation are eligible.
  * Unique to Europe (EU): Only participants who have pre-existing local results can be enrolled.
* For the ASP5834 monotherapy dose escalation part, participant with any histologically confirmed locally advanced (unresectable) or metastatic solid tumor malignancy is eligible. Participant must have received prior standard therapy in the advanced setting, and the investigator does not see any further clinical benefit from continuing such therapy or the participant is ineligible to receive standard approved therapies.
* For the ASP5834 monotherapy dose expansion part, the following criteria apply:

  * [pancreatic ductal adenocarcinoma (PDAC) Expansion Cohort(s)] Participant has histologically confirmed locally advanced (unresectable) or metastatic PDAC.
  * [PDAC Expansion Cohort(s)] Participant has a documented KRAS G12V, G12D, G12C, G12R, G12A or G13D mutation determined by local testing.
  * [PDAC Expansion Cohort(s)] Participant must have received standard therapy in the advanced setting, including prior therapy with a gemcitabine-based or fluoropyrimidine-based regimen or is ineligible for these therapies.
  * [PDAC Expansion Cohort(s)] No more than 2 prior lines of systemic therapy are allowed in the advanced setting (note: maintenance therapy does not count as a separate line of therapy).
  * [PDAC Expansion Cohort(s)] For a participant who received prior neoadjuvant or adjuvant chemotherapy and had recurrence on or within 6 months of completion of therapy, the neoadjuvant or adjuvant chemotherapy should be counted as a regimen in the advanced setting.
  * [non-small cell lung cancer (NSCLC) Expansion Cohort(s)] Participant has histologically confirmed locally advanced (unresectable) or metastatic NSCLC.
  * [NSCLC Expansion Cohort(s)] Participant has a documented KRAS G12V, G12D, G12R, G12A or G13D mutation determined by local testing.
  * [NSCLC Expansion Cohort(s)] Participant must have received standard therapy in the advanced setting, including prior platinum-based chemotherapy and checkpoint inhibitor therapy or is ineligible for these therapies. Participants with known actionable genomic alterations (AGA) must have received prior therapy with an approved targeted therapy in accordance with local requirements.
  * [NSCLC Expansion Cohort(s)] For a participant who has received prior neoadjuvant or adjuvant therapy and had recurrence during or within 6 months of completion of therapy, the neoadjuvant or adjuvant therapy should be counted as a regimen in the advanced setting (for those who received perioperative therapy, the entire course should be counted as therapy in the advanced setting).
  * [NSCLC Expansion Cohort(s)] For a participant with a history of unresectable Stage III disease who received prior multi-modal therapy and had recurrence on or within 6 months of completion of therapy, the multi-modal therapy should be counted as a therapy in the advanced setting. If chemoradiation was followed by treatment with checkpoint inhibitor therapy without documented progression between chemoradiation and checkpoint inhibitor therapy, the entire treatment course should be counted as therapy in the advanced setting.
  * [Other Solid Tumor Expansion Cohort] Participant has a histologically confirmed locally advanced (unresectable) or metastatic solid tumor type other than PDAC, colorectal cancer (CRC) or NSCLC.
  * [Other Solid Tumor Expansion Cohort] Participant has a documented KRAS G12V, G12D, G12C, G12R, G12A or G13D mutation or KRAS amplification (copy number >/=4) determined by local testing.
  * [Other Solid Tumor Expansion Cohort] Participant must have received prior standard therapy in the advanced setting, and the investigator does not see any further clinical benefit from continuing such therapy or is ineligible to receive standard approved therapies.
* For ASP5834 combination therapy dose escalation and dose expansion parts, the following criteria apply:

  * [CRC Dose Escalation and Dose Expansion Parts] Participant has histologically confirmed locally advanced (unresectable) or metastatic adenocarcinoma of the colon or rectum.
  * [CRC Dose Escalation and Dose Expansion Parts] Participant has a documented KRAS G12V, G12D, G12C, G12R, G12A or G13D mutation determined by local testing.
  * [CRC Dose Escalation and Dose Expansion Parts] Participant must have received standard therapy in the advanced setting, including prior therapy with fluoropyrimidine, oxaliplatin and irinotecan and anti-vascular endothelial growth factor (VEGF) therapy or is ineligible for these therapies.
  * [CRC Dose Escalation and Dose Expansion Parts] For a participant who has received neoadjuvant or adjuvant chemotherapy and had recurrence during or within 6 months of completion of therapy, the neoadjuvant or adjuvant chemotherapy should be counted as a regimen in the advanced setting.
  * [CRC Dose Escalation and Dose Expansion Parts] Participant with microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) colorectal cancer (CRC) must have also received prior treatment with immune checkpoint inhibitors or is ineligible for these therapies.
* Participant consents to provide tumor specimen in a tissue block or unstained serial slides or a baseline tumor biopsy obtained after the last interventional treatment, but not more than 90 days prior to the start of study intervention. Participant also consents to provide a tumor biopsy during the treatment period as indicated in the schedules of assessments. If a participant cannot provide a tumor specimen or undergo a baseline tumor biopsy procedure no more than 90 days prior to the start of study intervention, contact the medical monitor. Submission of an archival tumor tissue specimen to the central laboratory in addition to the baseline specimen is highly encouraged.
* Participant has at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participant's adverse event (AEs) (excluding alopecia) from prior anti-cancer therapy have improved to Grade 1 or baseline at least 14 days prior to the start of study intervention. Persistent Grade 2 or higher toxicities from prior anti-cancer therapy that are considered clinically irreversible, may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and sponsor.
* Participant has adequate organ function as indicated by laboratory values (if a participant has received a recent blood transfusion, the laboratory tests must be obtained >/= 14 days after any blood transfusion).
* Female participant is not pregnant confirmed by pregnancy test and medical evaluation by interview, and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who has a negative urine or serum pregnancy test within 7 days prior to day 1 and agrees to follow the contraceptive guidance from the time of informed consent through at least 6 months after final investigational study intervention administration.
* Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 6 months after final investigational study intervention administration.
* Female participant must not donate ova starting at first administration of study intervention and throughout the investigational period and for 6 months after final investigational study intervention administration.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 3 months after final investigational study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 3 months after final investigational study intervention administration.
* Male participant must not donate sperm during the treatment period and for 3 months after final investigational study intervention administration.
* Participant agrees not to participate in another interventional study while receiving study intervention in the present study/participating in the present study.

Exclusion Criteria:

* Participant has symptomatic or untreated central nervous system (CNS) metastases. Participants with stable, asymptomatic and treated CNS metastases are eligible.
* Participant has leptomeningeal disease as a manifestation of the current malignancy.
* Participant has another prior malignancy active (i.e., requiring treatment or intervention) within the previous 2 years different from the primary malignancy for this study, except for local malignancies that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast, which are allowed.
* Participant with active hepatitis B (including acute hepatitis B virus (HBV) or chronic HBV) or hepatitis C virus (HCV) (Ribonucleic acid (RNA) detected by qualitative assay). HCV RNA testing is not required in participants with negative HCV antibody testing.
* Participant has a known history of human immunodeficiency virus (HIV) infection with Acquired Immune Deficiency Syndrome (AIDS) related complications. No HIV testing is required unless mandated by a local health authority.
* Participant has had a myocardial infarction or unstable angina within 6 months prior to the start of study intervention or currently has an uncontrolled illness including, but not limited to symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia (including but not limited to uncontrolled atrial fibrillation, recent restoration of rhythm after atrial fibrillation, clinically significant conduction disorder within 6 months prior to the start of study intervention, or ventricular arrhythmias), obligate use of a cardiac pacemaker, or long QT syndrome.
* Resting heart rate < 50 bpm at screening, unless clinically appropriate (e.g., well-conditioned participant) and deemed not clinically significant.
* Known family history of sudden cardiac death before 50 years of age.
* Hypokalemia that is not corrected to within the institutional normal range prior to first dose of study intervention.
* Participants with clinically significant electrolyte abnormalities (e.g., hypomagnesemia or hypocalcemia) that are not corrected to within the institutional normal range prior to first dose of study intervention.
* Participant has had major surgery within 4 weeks prior to first dose of study intervention.
* Participant has acute neurological events (e.g., intracranial or subarachnoid hemorrhage, stroke, intracranial trauma) within 6 months prior to the first dose of study intervention.
* Participant has received any radiotherapy (including stereotactic radiosurgery) within 14 days prior to the first dose of study intervention.
* Participant has received prior KRAS targeting agents (including but not limited to KRAS directed inhibitors, degraders, small interfering RNA [siRNA] therapies, vaccines and cellular therapies), with the following exceptions:

  * In the dose escalation part, a participant with PDAC or NSCLC who has received prior RMC-6236 or RMC-9805 or a participant with NSCLC who has received prior KRAS G12C inhibitors but no other KRAS targeting agents will be eligible.
* Participant has an active infection requiring any systemic anti-infectious agents within 14 days prior to study intervention.
* Participant is expected to require another form of anticancer therapy while on study treatment.
* Participant requires treatment with concomitant drugs that are strong or moderate inhibitors or inducers of Cytochrome P450 family 3 subfamily A (CYP3A).
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any condition that makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to the protocol specified study intervention(s) or any components of the formulation used.
* Participant has a corrected QT interval by Fridericia (QTcF) value (single electrocardiogram (ECG)) of > 450 msec (men) or > 470 msec (women) during screening.
* Participant has a left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram (ECHO) (or multigated acquisition (MUGA)) performed at screening.
* Participant with a known history of an acquired KRAS G12V, G12D, G12C, G12R, G12A or G13D mutation or KRAS amplification identified as a resistance mechanism to prior systemic therapy (note: if a participant has more than 1 relevant KRAS alteration [KRAS G12V, G12D, G12C, G12R, G12A or G13D mutation or KRAS amplification], only those with a known history of acquired resistance to all relevant KRAS alterations would be excluded). Participant will not be excluded if it is not known whether the KRAS alteration(s) were acquired as a resistance mechanism.
* UNIQUE to EU: Participant who is the subject of any legal protection measures under local legislation will not be allowed.
* [ASP5834 combination therapy] Participant had prior discontinuation of panitumumab treatment due to toxicity or intolerance of panitumumab.
* [ASP5834 combination therapy] Participant has a history of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) (Dose Escalation only) | Up to 21 days
  A DLT is defined as any Adverse Event (AE) which meets DLT criteria, not clearly due to the underlying disease or extraneous causes, that occurs within the DLT observation period.
Number of participants with Adverse Events (AEs) | Up to 40 months
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
Number of Participants with Serious Adverse Events (SAEs) | Up to 40 months
  An SAE is any untoward medical occurrence that at any dose either results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other medical situation.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 40 months
  Number of participants with potentially clinically significant laboratory values.
Number of Participants with Eye Exam abnormalities and/or Adverse Events (AEs) | Up to 39 months
  Number of participants with potentially clinically significant eye exam values.
Number of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to 39 months
  Number of participants with potentially clinically significant ECG values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to 40 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with echocardiogram (ECHO) abnormalities and/or adverse events (AEs) | Up to 39 months
  Number of participants with potentially clinically significant ECHO values.
Number of participants with multigated acquisition (MUGA) abnormalities and/or adverse events (AEs) | Up to 39 months
  Number of participants with potentially clinically significant MUGA values.
Number of Participants with Physical Examination (PE) abnormalities and/or AEs | Up to 40 months
  Number of participants with potentially clinically significant PE values.
Number of Participants at each grade of Eastern Cooperative Oncology Group (ECOG) performance status scores | Up to 40 months
  The ECOG scale will be used to assess performance status. Scores range from 0 (fully active) to 5 (dead). Negative change scores represent an improvement. Positive scores represent a decline in performance.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) of ASP5834 per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 45 months
  ORR is defined as the proportion of participants whose best overall response is a Complete Response (CR) or Partial Response (PR) per RECIST v1.1.
Duration of Response (DOR) of ASP5834 per RECIST v1.1 | Up to 45 months
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented progressive disease (PD) per RECIST v1.1 or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) of ASP5834 per RECIST v1.1 | Up to 45 months
  DCR is defined as the proportion of participants whose best overall response is CR, PR or stable disease (SD) per RECIST v1.1.
Progression Free Survival (PFS) per RECIST v1.1 | Up to 45 months
  PFS is defined as the time from the first dose of study intervention until the date of documented radiological disease progression by investigator per RECIST v1.1 or until death for any cause, whichever comes first.
Overall Survival (OS) | Up to 45 months
  OS is defined as the time from the first dose of study intervention until death due to any cause.
Pharmacokinetics (PK) of ASP5834 in plasma: area under the concentration-time curve at 24 hours (AUC24h) | Up to 39 months
  AUC24h will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of ASP5834 in plasma: area under the concentration-time curve at 168 hours (AUC168h) | Up to 39 months
  AUC168h will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of ASP5834 in plasma: area under the concentration-time curve at 336 hours (AUC336h) for 1 of 2 dose regimens | Up to 39 months
  AUC336h will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of ASP5834 in plasma: maximum concentration (Cmax) | Up to 39 months
  Cmax will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of ASP5834 in plasma: trough concentration (Ctrough) | Up to 39 months
  Ctrough will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of ASP5834 in plasma: terminal elimination half-life (t1/2) | Up to 39 months
  t1/2 will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of ASP5834 in plasma: time of maximum concentration (tmax) | Up to 39 months
  tmax will be recorded from the PK plasma samples collected.
Change from baseline in Kirsten rat sarcoma viral oncogene homolog (KRAS) protein levels | Up to 45 months
  KRAS protein levels in tumor samples will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Lead, Study Director — Astellas Pharma Inc
Locations (11):
- United States (7):
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - START Midwest, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NEXT Oncology Dallas, Irving, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia
- France (2):
  - Site FR33003, Bordeaux, Nouvelle-Aquitaine
  - Site FR33001, Villejuif
- Spain (2):
  - Site ES34001, Madrid
  - Site ES34003, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as compounds terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency